CLINICAL TRIAL: NCT06031597
Title: Radiotherapy Combined With Immune Checkpoint Inhibitors (ICIs) as Treatment for Locally Advanced Non-small-cell Lung Cancer After Failing Induction Immuno-chemotherapy: a Prospective, Real-world Cohort Study.
Brief Title: Radiotherapy Combined With ICIs as Treatment for LA-NSCLC After Failing Induction Immunochemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xu Yujin, MD, Chief Physician, Department of Thoracic Radiotherapy, Zhejiang Cancer Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-700(IIT)
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer Stage III
Keywords: Non-small cell lung cancer; Immune checkpoint inhibitors; Radiotherapy; Radiation pneumonitis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Pneumonitis | interventions — Radiotherapy; Cisplatin; Immunotherapy; Nivolumab; atezolizumab; durvalumab; pembrolizumab; tislelizumab; sugemalimab; sintilimab; camrelizumab; Adjuvants, Immunologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A: concurrent chemoradiotherapy combined with ICIs (Experimental): For performance status (PS)=0-1 and both lungs V20≤20%, mean lung dose (MLD)≤11 gray(Gy), then the patient should be treated with concurrent chemo-radiotherapy and immunotherapy, and immunotherapy should be given after chemo-radiotherapy to maintain up to 1 year. Participants eligible for enrollment will receive radiotherapy within 8 weeks of the end of chemotherapy combined with Immune checkpoint inhibitors (ICIs) at a radical prescribed dose of 60 Gy ± 10% at 2 Gy once daily for 5 days per week. The chemotherapy regimen will be cisplatin at a dose of 25 mg/m2 once a week for 5-6 cycles. Marketed programmed cell death 1 (PD-1) or programmed cell death L1 (PD-L1) inhibitors are chosen as immunotherapy agents. Immunotherapy will be given every 3 weeks, with no more than 3 cycles of immunotherapy during radiotherapy. The dosage is recommended according to the drug insert.
  Interventions: Radiation: radiotherapy; Drug: Platinum-Based Drug; Drug: Immunotherapy; Drug: Immunotherapeutic Agent
- Cohort B: concurrent radiotherapy combined with ICIs (Experimental): For PS=0-1 and 20%<both lungs V20≤25% or 11Gy<MLD≤13Gy, radiotherapy alone combined with concurrent immunotherapy, followed by immunotherapy up to 1 year. Participants eligible for enrollment will receive radiotherapy within 8 weeks of the end of chemotherapy combined with ICIs at a radical prescribed dose of 60 Gy ± 10% at 2 Gy once daily for 5 days per week. Marketed PD-1 or PD-L1 inhibitors are chosen as immunotherapy agents. Immunotherapy will be given every 3 weeks, with no more than 3 cycles of immunotherapy during radiotherapy. The dosage is recommended according to the drug insert.
  Interventions: Radiation: radiotherapy; Drug: Immunotherapy; Drug: Immunotherapeutic Agent
- Cohort C: radiotherapy (Experimental): For PS=2 or 25%<both lungs V20≤30% or 13Gy<MLD≤17Gy, radiotherapy alone, followed by immunotherapy for up to 1 year. Participants eligible for enrollment will receive radiotherapy within 8 weeks of the end of chemotherapy combined with ICIs at a radical prescribed dose of 60 Gy ± 10% at 2 Gy once daily for 5 days per week. Marketed PD-1 or PD-L1 inhibitors are chosen as immunotherapy agents. The dosage is recommended according to the drug insert.
  Interventions: Radiation: radiotherapy; Drug: Immunotherapeutic Agent

INTERVENTIONS:
Radiation: radiotherapy — Radiotherapy techniques: Volumetric-modulated arc therapy (VMAT) and image guided radiotherapy (IGRT).
  Radiotherapy dose: Radical prescription dose of 60 gray (Gy) ± 10%, 2 Gy per session, once a day, 5 days a week.
Drug: Platinum-Based Drug — Cisplatin 25 mg/m2 once per week for a total of 5-6 cycles. For participants who have not completed 4 cycles of conversion chemotherapy in combination with immunotherapy, the original chemotherapy regimen may also be used, with the total number of chemotherapy cycles not exceeding 6 cycles.
  Other Names: Cisplatin
  Arms: Cohort A: concurrent chemoradiotherapy combined with ICIs
Drug: Immunotherapy — Concurrent programmed cell death 1 (PD-1) or programmed cell death L1 (PD-L1) inhibitors every 3 weeks during radiotherapy and no more than 3 doses during the course of radiotherapy.
  Other Names: Nivolumab; Atezolizumab; Durvalumab; Pembrolizumab; Tislelizumab; Sugemalimab; Sintilimab; Camrelizumab
  Arms: Cohort A: concurrent chemoradiotherapy combined with ICIs; Cohort B: concurrent radiotherapy combined with ICIs
Drug: Immunotherapeutic Agent — All participants will be evaluated within 1-42 days after receiving radiation (chemotherapy). If disease progression does not occur, adjuvant therapy with a PD-1 or PD-L1 inhibitor is continued until disease progression up to 1 year.
  Other Names: Nivolumab; Atezolizumab; Durvalumab; Pembrolizumab; Tislelizumab; Sugemalimab; Sintilimab; Camrelizumab

SUMMARY:
Patients with stage III non-small-cell lung cancer initially evaluated as unresectable are selected for the program, who are remained unresectable after 2-4 cycles of conversion chemotherapy combined with immune checkpoint inhibitors. Investigators will stratify the treatment according to different performance status scores and radiotherapy plan bi-lung receptor volume to evaluate the safety and efficacy of immunotherapy followed by combined radiotherapy.

DETAILED DESCRIPTION:
This is a prospective, real-world cohort study, which aimed to evaluate the safety and efficacy of immunotherapy followed by combined radiotherapy. Participants will be selected and entered into three different cohorts according to different performance status(PS) scores and radiotherapy schedules based on the amount of bilateral lungs treated. Cohort A: PS=0-1 and bilateral lung V20≤20%, mean lung dose(MLD)≤11 gray(Gy), radiotherapy and immunotherapy, followed by immunotherapy for up to 1 year; Cohort B: PS=0-1 and 20%<bilateral lung V20≤25% or 11 Gy<MLD≤13 Gy, radiotherapy combined with immunotherapy, followed by immunotherapy for up to 1 year; Cohort C: PS=2 or 25%<bilateral V20≤30% and 3 Gy <MLD≤ 17 Gy, radiotherapy alone, followed by immunotherapy for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed non-small cell lung cancer
2. Presence of at least one measurable lesion according to RECIST 1.1 criteria
3. Classified as American Joint Committee on Cancer staging system, eighth edition (AJCC-8) Stage III, initially evaluated as unresectable and reevaluated as unresectable after 2-4 cycles of induction chemotherapy combined with immunotherapy
4. Age 18-75
5. Eastern Cooperative Oncology Group (ECOG) physical state score of 0-2
6. Patients with the pathologic type of adenocarcinoma should be negative for driver genes (EGFR, anaplastic lymphoma kinase, ROS1)
7. Serum hemoglobin ≥ 90 g/L, platelets ≥ 90 × 109/L, absolute neutrophil count ≥ 1.2 × 109/L
8. Serum creatinine ≤ 1.25 times upper limit of normal(ULN) or creatinine clearance ≥ 60 mL/min
9. Serum bilirubin ≤ 1.5 times ULN, (AST) and alanine aminotransferase aspartate aminotransferase (ALT) ≤ 2.5 times ULN, alkaline phosphatase ≤ 5 times ULN
10. Forced expiratory volume in one second (FEV1)>0.8 liter
11. Normal coagulation function (Prothrombin time prolonged by no more than 3s and activated partial thromboplastin time prolonged by no more than 10s)
12. Patients signed a formal informed consent form to indicate that they understood that the study complied with the hospital's policies and ethical requirements

Exclusion Criteria:

1. The pathologic type is lung carcinoid or small cell lung cancer
2. Patients with any distant metastases
3. Grade 2 or higher unresolved toxic effects after conversion therapy (according to the Common Terminology Criteria for Adverse Events CTCAE)
4. A recent efficacy rating of PD after conversion therapy
5. Radiotherapy plan for normal lung tissue V20 > 30%, or average lung dose MLD > 17 Gy
6. Active or previous autoimmune disease (within the past 2 years) or history of primary immunodeficiency
7. Patients with any other previous or current malignancy, except non-melanoma skin or cervical cancer in situ
8. Any other disease or condition suggesting a contraindication to radiotherapy (e.g., active infection, within 6 months of myocardial infarction, symptomatic cardiac disease including unstable angina pectoris, congestive heart failure, or uncontrolled arrhythmias, immunosuppressive therapy)
9. Pregnant or nursing women
10. Women and men who are at risk of becoming pregnant but are unwilling to use adequate contraception
11. Evidence of hereditary bleeding disorders or coagulation disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
radiation pneumonitis | Within 6 months after radiation therapy
  Incidence of grade 2 or higher radiation pneumonitis.

SECONDARY OUTCOMES:
progression-free survival | 2 years
  Time from enrolment to disease progression or death from any cause or censored at the last follow-up.
overall survival | 3 years
  Time from enrolment to death or censored at the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Yujin, PhD, Study Director — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: No